CLINICAL TRIAL: NCT01423474
Title: Randomized Phase II Study of 2 Hypofractionated Radiotherapy Schedules for Low- and Intermediate-Risk Prostate Cancer
Brief Title: Prostate Accurately Targeted Radiotherapy Investigation of Overall Treatment Time
Acronym: PATRIOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CancerCare Manitoba (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Dr. Aldrich Ong, Radiation Oncologist, CancerCare Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 50-2011
Record Dates: First submitted 2011-08-23; First posted 2011-08-26 (Estimated); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Prostatic Neoplasms
Keywords: Radiotherapy; Hypofractionation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Image-Guided

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Short treatment time (11 days) (Experimental)
  Interventions: Radiation: Image-guided radiotherapy
- Long treatment time (29 days) (Experimental)
  Interventions: Radiation: Image-guided radiotherapy

INTERVENTIONS:
Radiation: Image-guided radiotherapy — 40 Gy / 5 fractions / 11 days
  Arms: Short treatment time (11 days)
Radiation: Image-guided radiotherapy — 40 Gy / 5 fractions / 29 days
  Arms: Long treatment time (29 days)

SUMMARY:
The purpose of this study is to compare the toxicity of two new radiation schedules for the treatment of prostate cancer. Patients will be randomized to receive 5 treatments delivered every other day over 11 days, or once per week over 29 days. Both of these schedules are shorter than the standard treatment which is usually 39 treatments over 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Low or intermediate risk prostate cancer patients as defined by:

  * Clinical stage T1-2b, Gleason Score <=7, and PSA <=20 ng/mL
* Age >= 18 years

Exclusion Criteria:

* Androgen deprivation therapy (LHRH-agonists or antiandrogens) >6 months
* Prior pelvic radiotherapy
* Anticoagulation medication (if unsafe to discontinue for gold seed insertion)
* Diagnosis of bleeding diathesis
* Large prostate (>90cm3) on imaging
* Immunosuppressive medications
* Inflammatory bowel disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Bowel related quality-of-life | 3 months

SECONDARY OUTCOMES:
Gastrointestinal toxicity | During radiotherapy, at 3 and 6 months, then every 6 months after
  Radiation Therapy Oncology Group Acute and Late Morbidity Scoring Schema
Genitourinary toxicity | During radiotherapy, at 3 and 6 months, then every 6 months after
  Radiation Therapy Oncology Group Acute and Late Morbidity Scoring Schema
PSA relapse rate | 3 and 5 years
Patient Overall Quality of life | During radiotherapy, at 3 and 6 months, then every 6 months after
Salvage androgen deprivation therapy rate | 3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Aldrich Ong, MD, Principal Investigator — CancerCare Manitoba; Andrew Loblaw, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (3):
- Canada (3):
  - BC Cancer Agency - Abbotsford Centre, Abbotsford, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ong WL, Quon H, Ong A, Cheung P, Chu W, Chung H, Vesprini D, Chowdhury A, Panjwani D, Alayed Y, Pang G, Korol R, Davidson M, Ravi A, McCurdy B, Zhang L, Kulasingham-Poon M, Mamedov A, Deabreu A, Loblaw A. Every Other Day or Once a Week: Long-term Oncological Outcomes in the Phase 2 PATRIOT Trial of Prostate Stereotactic Ablative Body Radiotherapy. Eur Urol Oncol. 2025 Aug;8(4):909-913. doi: 10.1016/j.euo.2025.03.011. Epub 2025 Apr 26. PMID 40288917
- [Derived] Quon HC, Ong A, Cheung P, Chu W, Chung HT, Vesprini D, Chowdhury A, Panjwani D, Pang G, Korol R, Davidson M, Ravi A, McCurdy B, Zhang L, Mamedov A, Deabreu A, Loblaw A. Once-weekly versus every-other-day stereotactic body radiotherapy in patients with prostate cancer (PATRIOT): A phase 2 randomized trial. Radiother Oncol. 2018 May;127(2):206-212. doi: 10.1016/j.radonc.2018.02.029. Epub 2018 Mar 15. PMID 29551231